CLINICAL TRIAL: NCT03715920
Title: Comparison of Different Quadriceps Femoris Isometric Strengthening Methods in Healthy Young Women
Brief Title: Comparison of Different Quadriceps Femoris Isometric Strengthening Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bilge Basakci Calik, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 60116787-020/77612
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Muscle Strength
Keywords: Quadriceps femoris; isometric form; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy; Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Voltage Pulsed Galvanic Current (Active Comparator): HVPG current is a new form of neuromuscular electrical stimulation.The total output voltage of the device ranged from 0 to 500 volts and the current intensity was increased until the sensible contraction of the applied muscle was achieved without causing too much sense of discomfort
  Interventions: Device: Electrical currents
- Russian Current (Placebo Comparator): Russian currents are a high frequency current of 2500 Hz and reduce the resistance of the skin and it would penetrate deeper and reach deeper motor nerves.Russian movement, a protocol developed by Kots, also known as "Russian Technique", was used in the literature. There were 10 muscle contractions per treatment session in this protocol. Each contraction lasted for 10 seconds and a resting time of 50 seconds were given for the next contraction (transition: rest ratio was 1/5).
  Interventions: Device: Electrical currents
- Isometric Exercise (Sham Comparator): Isometric or static strength training is exercises performed without joint movement and changing muscle length during muscle contraction.
  The body and knee of the participants in the isometric exercise group were positioned and stabilized at 75 ° flexion and 60 ° flexion angle, respectively as in the stimulation groups. Participants were asked to do 10 repetitions as 10 seconds of maximum voluntary contractions and 10 seconds of rest.
  Interventions: Device: Electrical currents

INTERVENTIONS:
Device: Electrical currents — The training was planned as HVPG current for the the first group (n = 16), as Russian current for the second group (n = 15) and as isometric strengthening for the third group (n = 15). All treatments were performed under physiotherapist supervision for a total of 15 sessions for 3 days a week for 5 weeks.
  Other Names: Exercises; Isometric

SUMMARY:
Background:It has been reported in previous studies that more motor units are fired with electrical stimulation than voluntary muscle contraction, and even high intensity currents provide 10-30% more contractions than voluntary muscle contraction.

Objective:This study was planned to compare the effectiveness of high voltage pulsed galvanic (HVPG) stimulation, Russian current and isometric exercise on quadriceps femoris (QF) isometric muscle strength in healthy young women.

Methods:Forty-six healthy young women were included in the study (mean age=21.02 ± 1.27). Before and after the training, the dominant side QF isometric muscle strength of participants was assessed with the Isokinetic Dynamometer . The peak torque and average torques of the participants were recorded after the test. The training was planned as HVPG current for the the first group (n = 16), as Russian current for the second group (n = 15) and as isometric strengthening for the third group (n = 15). All treatments were performed under physiotherapist supervision for a total of 15 sessions for 3 days a week for 5 weeks.

DETAILED DESCRIPTION:
Muscle strength, Isokinetic strength measurement:

The dominant side QF isometric muscle strength (torque measurements) of the participants was assessed with the Isokinetic Dynamometer . Before the test, participants were subjected to a standard warm-up of 5 minutes and evaluations were carried out using a standard seat. The back of the seat was angled 105 ° backward to provide 75 ° flexion at the body. The knee was positioned at an angle of 60 ° and was fixed with bands around the body, waist, hip and ankle. Participants had no previous experience with isokinetic dynamometer testing, therefore; it was started with a trial whose protocols were same with QF isometric muscle strength measurement protocols. Then participants QF isometric muscle strength was measured by three 10-second maximal isometric contraction. Rest periods of 3 seconds between each contraction were given. Each participant held the sides of the seat with both hands during the test. Verbal encouragement was made throughout the whole test to obtain maximum strength from the participants. The peak torque and average torques of the participants were recorded after the test.

High Voltage Pulsed Galvanic Current:

The instrument was automatically set to a pulse rate of 100 μs while the pulse frequency was set to 60 pulses / sec. In order to avoid fatigue, the intermittant form of the current was selected and the transition time / rest time was set to 4 sec. impulse / 12 sec. The total output voltage of the device ranged from 0 to 500 volts and the current intensity was increased until the sensible contraction of the applied muscle was achieved without causing too much sense of discomfort. Stimulation was performed after the body and knee were positioned and stabilized at 75 ° flexion and 60 ° flexion angle, respectively. One of the 6 * 8 cm carbonated electrodes was placed in the distal portion of the vastus medialis, while the other one was placed in the proximal portion of the vastus lateralis. This placement was intended to stimulate a large proportion of the muscle fibers of the QF muscle.The HVPG was applied for a total of 20 minutes. Current intensity was increased to obtain optimal muscle contraction.

Russian Current In the treatment with the Russian current, a protocol developed by Kots, also known in the literature as "Russian Technique", was used. In the treatment with the Russian movement, a protocol developed by Kots, also known as "Russian Technique", was used in the literature. There were 10 muscle contractions per treatment session in this protocol. Each contraction lasted for 10 seconds and a resting time of 50 seconds were given for the next contraction (transition: rest ratio was 1/5).The position of the participants in the application and the placement of the electrodes were same as the the other application. Current intensity was increased until tetanic muscle contraction was obtained.

Isometric Exercise:

The body and knee of the participants in the isometric exercise group were positioned and stabilized at 75 ° flexion and 60 ° flexion angle, respectively as in the stimulation groups. Participants were asked to do 10 repetitions as 10 seconds of maximum voluntary contractions and 10 seconds of rest.

ELIGIBILITY:
Inclusion Criteria:- Willingness to participate in the study.

* Not having knee complaints such as pain, lockout, morning arrest, swelling, difficulty in walking.
* Not having any orthopedic or neurological disability

Exclusion Criteria:

* Exercising regularly for the last six months.
* Presence of cardiovascular, pulmonary, orthopedic and neurological problems which may prevent exercise.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-24 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Isokinetic Strength measurement | One week
  Muscle strength, Isokinetic strength measurement:
  The dominant side QF isometric muscle strength (torque measurements) of the participants was assessed with the Isokinetic Dynamometer (Humac Norm Testing Rehabilitation System, CSMI Medical Solutions, USA).

SECONDARY OUTCOMES:
Isometric exercise | One week
  The body and knee of the participants in the isometric exercise group were positioned and stabilized at 75 ° flexion and 60 ° flexion angle, respectively as in the stimulation groups

CONTACTS AND LOCATIONS:
Locations (1):
- Bilge Basakci Calik, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03715920/Prot_000.pdf